CLINICAL TRIAL: NCT05221385
Title: A Phase Ia, Open-label, Dose Escalation Study of Safety, Tolerability, Pharmacokinetics of Gentulizumab, an Anti-CD47 Monoclonal Antibody, in Patients With Advanced Solid Malignancies and Non-Hodgkin Lymphoma (NHL)
Brief Title: Gentulizumab in Patients With Advanced Solid Malignancies and Non-Hodgkin Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to changes in the sponsor's research strategy
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Gensci059-Ia-A
Record Dates: First submitted 2021-12-27; First posted 2022-02-03 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Solid Tumor; Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental cohort (Experimental): Gentulizumab monotherapy 0.1, 0.3, 1, 3, 10, 30, 45 mg/kg administered intravenously once every week.
  Interventions: Drug: Gentulizumab

INTERVENTIONS:
Drug: Gentulizumab — Gentulizumab is administered IV once a week, with every 4 weeks as an administration cycle.

SUMMARY:
The purpose of this study is to assess the safety and tolerability of gentulizumab, an anti-CD47 Monoclonal Antibody, in participants with solid tumors and non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
This is a first-in-human, escalating dose trial of an antibody that inhibits an anti-apoptotic signal in human macrophages. The major aims of the study are to define the safety profile of this new drug, and to determine a recommended dose and schedule for potential additional trials.

ELIGIBILITY:
Inclusion Criteria:

* The patient has the willingness to communicate with the investigator, can understand and follow the trial requirements, is willing to participate in the trial, understands and signs a written Informed Consent Form（ICF）, and is willing and able to comply with the visit schedule, administration plan, laboratory examination, and other clinical trial procedures.
* Gender: Male or female.
* Age 18-70 years old.
* Expected survival ≥ 12 weeks.
* Patients with Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Patients with advanced solid tumors or NHL by histopathological diagnosis do not have acceptable standard treatment currently.
* Adequate organ function per protocol-defined criteria.

Exclusion Criteria:

* Use of protocol-defined prior/concomitant therapy.
* Currently receiving or has received an investigational treatment as part of a study within 4 weeks before the first dosing.
* History of severe hypersensitivity reaction to study treatments or their excipients.
* Known active central nervous system metastases.
* History of any active autoimmune disease history, or disease or syndrome requiring treatment with systemic steroids or immunosuppressive medications.
* Presence of active infection.
* Known additional malignancy that has not been cured in the last 5 years.
* Any uncontrolled intercurrent illness or condition that in the judgment of the Investigator may endanger the patient.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of Gentulizumab as Measured by the Number of Participants Experiencing Dose-limiting Toxicities (DLTs), Adverse Events (AEs), and Serious Adverse Events (SAEs). | 28 days
  The CTCAE criteria will be used to assess adverse events on this trial.
Pharmacokinetic (PK) Parameter: Area under the plasma concentration versus time curve (AUC). | From the first dosing to 90 days after the last dosing
Pharmacokinetic (PK) Parameter: Peak plasma concentration (Cmax). | From the first dosing to 90 days after the last dosing
Pharmacokinetic (PK) Parameter: Terminal phase half-life (t1/2). | From the first dosing to 90 days after the last dosing

SECONDARY OUTCOMES:
Pharmacodynamic (PD) Characteristics of Gentulizumab. | From the first dosing to 90 days after the last dosing
  PD parameters include: receptor occupancy (RO) of gentulizumab of red blood cells, and white blood cells in peripheral blood.
Immunogenicity of Gentulizumab. | From the first dosing to 28 days after the last dosing
  Numbers of anti-drug antibody (ADA) and/or neutralizing antibody (NAb) positive participants will be used to assess the immunogenicity of gentulizumab.

OTHER OUTCOMES:
Objective Response Rate (ORR) of Gentulizumab as Monotherapy. | From date of first dosing until the date of disease progression or death due to any cause, whichever came first, assessed up to 12 months.
  ORR was defined as the percentage of participants who had complete response (CR) or partial response (PR) per RECIST v1.1 by investigator determination.
Progression-free Survival (PFS) of Gentulizumab as Monotherapy. | From date of first dosing until the date of disease progression or death due to any cause, whichever came first, assessed up to 12 months.
  PFS was defined as the time ranging from the beginning of enrollment to the tumor progression for the first time or death.
Exploratory indicators related to biomarkers | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhang, Doctor, Principal Investigator — Fudan University
Locations (2):
- China (2):
  - Jian Zhang, Shanghai, Shanghai Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No